CLINICAL TRIAL: NCT05402254
Title: Evaluation of the Impact of a Pharmacovigilance Program Led by Advanced Practice Nursing on Patients and Professionals at Hospital: Intervention Study
Brief Title: Impact of a Pharmacovigilance Program Led by Advanced Practice Nursing
Acronym: IMPACTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natalia Rodriguez Galan (Other)
Responsible Party: Sponsor-Investigator, Natalia Rodriguez Galan, principal investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EI-FC-2022-03
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Adverse Drug Event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacovigilance Program (Experimental): Intensive nursing intervention is carried out for the identification and notification of ADE
  Interventions: Other: Pharmacovigilance Program
- Control (No Intervention): The Usual practice of the nursing care process

INTERVENTIONS:
Other: Pharmacovigilance Program — Knowledge of the risks in the use of the drug, identification and notification of ADE
  Arms: Pharmacovigilance Program

SUMMARY:
HYPOTHESIS An advanced practice nursing intervention in the area of pharmacovigilance performed on patients and professionals improves the identification and reporting of suspected adverse drug reactions (ADR) and improves the overall experience of hospitalized patients.

DETAILED DESCRIPTION:
PRIMARY OBJETIVES

1. To assess whether an advanced nursing intervention improves the identification and reporting of suspected ADR.

SECONDARY OBJECTIVES

1. To determine if an advanced nursing intervention improves the experience related to the use of medications measured through the QExPac-21 patient experience questionnaire.
2. Identify which factors associated with medications increase the risk of ADRs and the characteristics of the patients.
3. Know the incidence and describe ADRs: severity, preventability, and causality using validated scales.
4. Describe the degree of nursing intervention according to the North American Nursing Diagnosis Association (NANDA) Taxonomy, and the classification of nursing interventions (NIC) Related to drug use.
5. Quantify the number of interconsultation generated by patients and professionals related to the use of drugs.
6. Determine the degree of adherence and compliance with the regimens prescribed to the patients.

STUDY DESIGN Prospective, randomized and controlled study of an intervention that compares a group of patients according to the usual practice of the nursing care process, against another on which a more intensive nursing intervention is carried out for the identification and notification of ADRs. It is carried out on a representative sample of patients admitted to a tertiary level hospital with 860 beds of the Madrid Health Service during the year 2022.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pharmacological treatment.
2. Patients of both sexes aged between 0 and 100 years.
3. Patients admitted to medical or surgical hospitalization units or emergency services for at least 24 hours.
4. Patients who have received the information and agreed to participate in the study.

Exclusion Criteria:

1. Patients included in other clinical trials or drug studies at the time of selection.
2. Patients with significant cognitive impairment, without adequate family support or primary caregiver.
3. Patients and/or caregivers who, once offered to participate in the study, do not give their consent
4. Impossibility of communication due to language barriers or other biopsychosocial problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Adverse drug event | Seven months
  Number of identified adverse drug event

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rodriguez Galán, Principal Investigator — Hospital San Carlos
Locations (1):
- Hospital San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No